CLINICAL TRIAL: NCT03512782
Title: Effectiveness of the Monitoring of Signs and Symptoms After Discharge From Hospital of Patients With Heart Failure
Brief Title: Post-discharge Monitoring of Patients With Heart Failure
Acronym: CARDIOENF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5085_15
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (No Intervention)
- INTERVENTION (Experimental)
  Interventions: Other: CARDIOENF

INTERVENTIONS:
Other: CARDIOENF — The patients listed in interventional group will have access to software Cardioenf that is a app used in a device (cel phone, tablet) to monitoring signs and symptoms of the heart failure patients after discharge from hospital. In this software, their signs and symptoms will be inserted in three moments during the first 30 days after discharge. Nurses will monitor these data in the follow-up period.
  Arms: INTERVENTION

SUMMARY:
What is proposed in this project is to develop and evaluate the effectiveness of an online remote monitoring system that is easily accessible to patients so that professionals with experience in monitoring patients with heart failure (HF) can monitor signs and symptoms of decompensation of the disease, as well as self-care actions. A randomized, blind trial for outcome evaluation was designed that will include patients hospitalized for acute HF at a referral institution in cardiology in southern Brazil. Patients in the intervention group will be followed up with a remote monitoring system, accessible by device (computer, tablet and cell phone) connected to the internet, by checking for signs, symptoms and self-care actions in three moments during 30 days after hospital discharge. Patients in the control group will follow up according to the routine of the hospital or physician assistant. The primary endpoint for assessing the efficacy of the system will be hospital readmission within 30 days (follow-up period). The information regarding the signs, symptoms and self-care of the patients will be monitored by the research team through an access schedule. The sample calculation points to the need to include a total of 142 patients (71 in each group). The data will be analyzed through descriptive and analytical statistics. It is hoped that the development of a remote monitoring system could be characterized as a strategy for the early detection of signs and symptoms of acute decompensation in HF patients, impacting on hospital readmission rates within 30 days after discharge. In addition, remote monitoring of signs and symptoms may promote improved adherence and self-care of patients. The scientific contribution will occur to the extent to which there is innovation in patient follow-up and feedback obtained from the patient's interaction with the system.

ELIGIBILITY:
Inclusion Criteria:

* with diagnosis of HF or hospitalized for acute HF

Exclusion Criteria:

* degenerative neurological diseases;
* patients with renal / hepatic / pulmonary or systemic disease that may confuse the interpretation of findings or result in limited life expectancy;
* surgical or therapeutic plan that may influence the follow-up;
* pregnancy;
* diagnosis of acute HF secondary to: sepsis, myocarditis, acute myocardial infarction, peripartum and other acute cause;
* not be able to contact by phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
hospital readmission | 1 month
  admission to the emergency department or hospitalization

SECONDARY OUTCOMES:
signs and symptoms of decompensation of heart failure | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Ciências da Saúde de Porto Alegre (UFCSPA), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No